CLINICAL TRIAL: NCT05842642
Title: Effects of Adding an Oculomotor Therapy Treatment to a Cervical Protocol in Patients With Migraine
Brief Title: Effects of Adding an Oculomotor Therapy Treatment in Patients With Migraine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Jaén (Other)
Responsible Party: Principal Investigator, Alexander Achalandabaso, Clinical Professor, University of Jaén
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Universidad de Alcalá
Record Dates: First submitted 2023-02-07; First posted 2023-05-06 (Actual); Last update posted 2023-09-18 (Actual); Status verified 2023-09

CONDITIONS: Migraine
Keywords: migraine; oculomotor; manual therapy; cervical
MeSH Terms: conditions — Migraine Disorders | interventions — SETX protein, human

STUDY DESIGN:
Intervention Model Description: Two groups, a control group and an experimental group. In the control group, a treatment of the cervical region will be done for 6 weeks, once a week, and they will be taught some exercises to do at home. And in the experimental group, the treatment of the control group will be done plus an additional intervention in the oculomotor region together with some specific exercises.
Who Masked: Participant
Masking Description: Upon acceptance, each participant will be assigned a treatment group. Before starting the intervention, all the subjects will go to the UAH physiotherapy center for a first visit with the first examiner where personal data will be collected and sociodemographic, psychometric and functional variables will be assessed.
  At the end of said evaluation, a second examiner gave them the steps to follow to carry out the study. In addition, you will be given a document with a table that will be your migraine diary that you must fill in every day from the start of treatment until the day of the last assessment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cervical treatment (Placebo Comparator): A treatment of the cervical region will be done for 6 weeks, once a week, and they will be taught exercises to do at home.
  Interventions: Other: Cervical
- Oculomotor treatment (Experimental): An oculomotor treatment will be added to the treatment of the cervical group with specific exercises in the area. Once a week during 6 weeks
  Interventions: Other: Cervical; Other: Oculomotor

INTERVENTIONS:
Other: Cervical — 6 weeks of treatment
Other: Oculomotor — 6 weeks of treatment
  Arms: Oculomotor treatment

SUMMARY:
Headaches are the fourth cause/reason for disability in the world population. Of which, headache in general accounts for 47%, 38% are tension headaches, 10% migraines and 3% for chronic headache lasting more than 15 days a month.

Migraine is a neurological disease/disorder originating in the central nervous system with difficulty modulating responses to common sensory stimuli.

Different studies have linked possible oculomotor problems and headaches, being an important and complex relationship.

It is difficult to find a suitable and beneficial treatment for the treatment of migraine. It is hypothesized that adding a treatment of manual therapy and therapeutic exercise of the oculomotor system to an already established protocol of manual therapy and therapeutic exercise of the cervical region, has an additional benefit for patients with migraines (in relation to the quality of life, symptomatology and functionality).

DETAILED DESCRIPTION:
Migraine is a neurological disease/disorder originating in the central nervous system with difficulty modulating responses to common sensory stimuli. It is characterized by being unilateral, frontotemporal, pulsatile, of moderate or severe intensity, nausea and/or vomiting, sensitivity to movement, visual, auditory, and other afferent stimuli may appear. In addition, other symptoms such as fatigue, neck stiffness, decreased concentration, mood swings and yawning may appear, and the headache may be anticipated up to 48 hours.

It has been hypothesized that the possible relationship between the eyes and the pathophysiology of migraine is due to the trigeminal-cervical complex, since if there is an alteration it would be established by a nociceptive impulse that can trigger central sensitization in the trigeminal nuclei.

Today, the quintessential treatment is pharmacological where the excessive use of medications can trigger possible side effects such as depression, anxiety, weight gain, fatigue and drowsiness, among others, causing an alteration in the patient's quality of life more than of the migraine attack.

Several studies show that there are other non-pharmacological treatment options such as manual physiotherapy and therapeutic exercise for migraines, and that it is effective for reducing the intensity and frequency of attacks, the use of medication and improving the quality of life. Being preventive treatments in order to avoid the frequency and intensity of these attacks.

At present, the role of oculomotricity in headache, although it may be promising, has not been extensively studied. In the literature that the investigators have reviewed, the investigators have found very few studies that investigate manual therapy directly on the eyeball, despite the great relationship of the trigeminal-vascular nerve with migraines and how it influences the different variables.

The main objective of the present study is to investigate the impact and possible additional benefits of adding an oculomotor treatment to a manual therapy protocol of the cervical region in patients with migraine.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18-65 years
* Suffer less than 15 days of headache per month,
* The pain must have these characteristics: unilateral, pulsating, of moderate to severe intensity, during the attack, nausea and/or vomiting, with the possible presence of an aura
* History of evolution of more than a year,
* Onset and aggravation in the afternoon and
* Relation to visual work
* Feeling of eye discomfort,
* Photophobia
* Neck pain after attack.

Exclusion Criteria:

* Receiving some type of preventive physiotherapy treatment at the time of the intervention
* Subjects with preventive medication, pregnancy or lactation, with neurological, systemic or psychiatric disorders, suffering from bone degeneration
* Metabolic or musculoskeletal problems that could imply risk of the vertebral artery
* Dizziness
* Unbalanced tension
* Use of specific medication
* Lack of fluency in Spanish.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2023-04-03 (Actual); Primary Completion 2023-05-30 (Actual); Study Completion 2023-09-15 (Actual)

PRIMARY OUTCOMES:
Changes in the impact | Baseline, 6 weeks and 3 months after intervention
  Using the Headache Impact Test (HIT-6) Questionnaire

SECONDARY OUTCOMES:
Changes in the pain | Baseline, 6 weeks and 3 months after intervention
  Using the Visual Analog Scale (VAS). Each item is scored 0-10 (0= no pain; 10= the major pain that the patient can imagine) yielding a total between 0 and 10.
Changes in the disability | Baseline, 6 weeks and 3 months after intervention
  Using the Migraine Disability Assessment (MIDAS) Questionnaire
Changes in the depression | Baseline, 6 weeks and 3 months after intervention
  Using the Patient Health Questionnaire (PHQ-9) Questionnaire
Changes in the anxiety | Baseline, 6 weeks and 3 months after intervention
  Using the Generalized Anxiety Disorder (GAD-7) Questionnaire
Changes in the sleep quality | Baseline, 6 weeks and 3 months after intervention
  Using the Pittsburgh Sleep Quality Index (PSQI) Questionnaire
Changes in the kinesiophobia | Baseline, 6 weeks and 3 months after intervention
  Using the Tampa Scale of Kinesiophobia (TSK-11) Questionnaire
Changes in the catastrophizing | Baseline, 6 weeks and 3 months after intervention
  Using the Pain Catastrophizing Scale (PCS) Questionnaire
Changes in the central sensitization | Baseline, 6 weeks and 3 months after intervention
  Using the Central Sensitization Inventory (CSI) Questionnaire
Changes in the neck disability | Baseline, 6 weeks and 3 months after intervention
  Using the Neck Disability Index (NDI) Questionnaire
Changes in the head repositioning | Baseline, 6 weeks and 3 months after intervention
  Using the Head Repositioning. This test will be used to assess the subject's proprioceptive ability to reposition the head on the trunk in the horizontal and sagittal planes and to measure the impact of treatment techniques.
  The distance between the center of the objective (target) and the laser point is measured, representing the cervico-cephalic positioning error
Changes in the strength of the deep cervical flexors | Baseline, 6 weeks and 3 months after intervention
  Using the Grimmer Test
Changes in the ocular movement | Baseline, 6 weeks and 3 months after intervention
  Using Smooth tracking test. It consists of following with the eyes an object (stick with a painted dot) that moves in the shape of an "H".
Changes in the ocular movement with variation of the head | Baseline, 6 weeks and 3 months after intervention
  Using the Smooth Pursuit Neck Torsion. It consists of following with the eyes an object (stick with a painted dot) that moves in the shape of an "H" with variant head position
Changes in the range of movement | Baseline, 6 weeks and 3 months after intervention
  Using the Cervical Range of Motion Instrument
Changes in the quality of life | Baseline, 6 weeks and 3 months after intervention
  Using the Short-Form 12 Health Survey (SF-12). Composed of twelve items, eight dimensions (physical function, physical role, bodily pain, mental health, general health, vitality, social function, and emotional role). The score ranges from 0 to 100, where the higher score implies a better health-related quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Achalandabaso, PhD, Study Director — University of Jaen
Locations (1):
- Physiotherapy clinic, Madrid, Spain